CLINICAL TRIAL: NCT04454333
Title: COVID-19 in Pain Perspective
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2811
Record Dates: First submitted 2020-06-30; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Infection; COVID; Pain
Keywords: infections; pain; Coronavirus
MeSH Terms: conditions — Infections; Pain; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized caused by COVID-19: A total of 466 patients hospitalized with the diagnosis of SARS-COV-2 at the University of Health Sciences, Şişli Hamidiye Etfal Training and Research Hospital were retrospectively screened. 212 of these patients did not answer the calls, 34 of them could not be reached because they gave the wrong phone number beforehand. 4 of the patients called by the phone had communication problems due to language problems and 10 people did not want to fill the questionnaire. 206 of them were contacted by the phone and their pain and myalgia in the head, neck-back, waist, shoulder and hip regions before, during and after SARS-COV-2, their anxiety and depression levels after SARS-COV-2, and their quality of life were questioned.

SUMMARY:
In our hospital's Infectious Diseases and Clinical Microbiology service, patients who have been hospitalized due to Covid -19 infection have a musculoskeletal pain and headache during this process, and 466 patients will be recruited to compare them with the pre-disease state of the patients and to evaluate the pain status of the patients after treatment.

DETAILED DESCRIPTION:
This retrospectively designed study was carried out by analyzing SARS-CoV-2 infected and hospitalized patients in our hospital for 2 month. The patients, whose contact information can be accessed from the hospital records, will be called by phone and pain inquiries were made during the SARS-CoV-2 infection process. In addition, patients' demographic data, living conditions (number and characteristics of the person in the household), comorbidities, symptom inquiry related to infection, duration of symptoms, length of hospitalstay, pre-infection pain conditions and current pain, anxiety, depression levels and quality of life will be questioned.

The pain questioning include the painful body region/s, severity (Numeric Rating Scale), type of analgesic drugs used, and duration of use that occurred during infection. Anxiety and depression levels will be evaluated, hospital anxiety and depression scale (HADS), and quality of life will be evaluated with SF-12 health assessment questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive PCR test results obtained from combined throat and nasopharyngeal swab samples
* patients consistent with Covid-19 infection as a result of thorax computed tomography, although PCR test results were negative.

Exclusion Criteria:

* Patients who have undergone surgery and trauma in the painful area in the past 3 months,
* Patients with pathological disease that can cause underlying pain
* Pregnant women
* Those who have psychiatric illness and use psychiatric drugs
* Presence of malignancy
* Patients with severe cognitive deficits

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our hospital, patients who were treated with the diagnosis of COVID-19 were selected. During the selection, patients between the ages of 18-95 were selected, considering the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale for Pain | up to 10 weeks
  Evaluation of severity of pain for head, back-neck and extremities by Numeric Rating Scale. Scoring will be done between 0 minimum and 10 maximum values. Higher scores mean worse outcome.
Hospital Anxiety and Depression Scale (HADS) | up to 10 weeks
  Evaluation of patient's anxiety and depression level in hospital by Hospital Anxiety and Depression Scale (HADS). The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report screening scale. It contains two 7-item scales: one for anxiety and one for depression both with a score range of 0-21. Higher scores mean a worse outcome.
SF-12 Health assesment Questionaire | up to 10 weeks
  Evaluation of patient's quality of life by SF-12 Health assesment Questionaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Ayyıldız, MD, Principal Investigator — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Sahin T, Ayyildiz A, Gencer-Atalay K, Akgun C, Ozdemir HM, Kuran B. Pain Symptoms in COVID-19. Am J Phys Med Rehabil. 2021 Apr 1;100(4):307-312. doi: 10.1097/PHM.0000000000001699. PMID 33480608